CLINICAL TRIAL: NCT01025908
Title: Cognitive-behavioural Therapyin Panic Disorder: the Preparation of Patients With Panic Disorder for Interoceptive and in Vivo Agoraphobic Exposure
Brief Title: Cognitive Behavior Psychotherapy in Panic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Antonio Egidio Nardi, Institute of Psychiatry - Federal University of Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LABPR
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2010-02-01 (Estimated); Status verified 2009-12

CONDITIONS: Panic Disorder; Agoraphobia
Keywords: psychotherapy; panic disorder; anxiety; behavior; cognition
MeSH Terms: conditions — Panic Disorder; Agoraphobia; Anxiety Disorders; Behavior | interventions — Psychotherapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): 25 panic disorder patients
  Interventions: Behavioral: Psychotherapy
- Supportive psychotherapy (Active Comparator): 25 panic disorder agoraphobia
  Interventions: Behavioral: Supportative psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy — Cognitive Behavioral Therapy
  Other Names: Cognitive Behavior psychotherapy
  Arms: Cognitive Behavioral Therapy
Behavioral: Supportative psychotherapy — Supportative psychotherapy
  Other Names: non-specific psychotherapy
  Arms: Supportive psychotherapy

SUMMARY:
The objective of this study in cognitive-behavioural therapy (CBT) was to demonstrate the preparation of the patient with panic disorder for agoraphobic exposures. The focus of the work consisted of interoceptive exposures, in vivo, of body sensations themselves, to feared places and situations. The sample consisted of 50 individuals. Group 1 undertook 10 weekly, individual sessions of CBT of one hour duration. Group 2, control, was just follow-up with supportive therapy. The procedures used for the exposures, especially for induction symptom exercises, were considered essential in the preparation of patients with panic disorder, to be able to face up to panic attacks and subsequent agoraphobic situations.

DETAILED DESCRIPTION:
The patients with PDA were diagnosed by medical psychiatrists from the team at the Respiration and Panic Laboratory of Instituto de Psiquiatria da Universidade Federal do Rio de Janeiro (IPUB/UFRJ), INCT Translational Medicine, according to the criteria of diagnostic of the Manual of Diagnostic and Statistics of Mental Disorder (DSM-IV-TR, 2002b) and according to the evaluation instrument SCID-I (Structured Clinical Interview Diagnostic) (First et al, 1997). The sample consisted of 50 voluntary patients divided in two Groups. The 1st Group, made up of 25 individuals, received 10 sessions of CBT. The 2nd Group, "control", also consisted of 25 patients, who received just supportive psychotherapy.

With a view to comparing the results of the Groups after the interventions, the following evaluation instruments were applied at the beginning and at the end of the research: Beck Anxiety Inventory (Beck et al, 1998a); State-Trait Anxiety Inventory (Spielberg et al, 1970); Sheehan Disability Scale (Sheeham, 1983a); Global Assessment of Functioning (AXIS V) (DSM-IV-TR, 2002c); questionnaire of fears and phobias (Mark & Mathews, 1979); questionnaire of cognitive agoraphobias( Chambless, 1984a); questionnaire of body sensations (Chambless, 1984b) and Panic and Agoraphobia Scale (Bandelow, 1999a).

The criteria for inclusion in the research was patients over 18 years old of both sexes with a diagnosis of PDA, with no serious comorbidities. The patients that presented alcohol or drug dependency, mental retardation or serious mental disorders were excluded from the research.

The patients who agreed to participate in the study, signed a "Term of Free and Clarified Consent" and were made aware of all the procedures undertaken, approved by the Committee of Ethics for the research IPUB/UFRJ.

In the evaluation of the tests the Chi-square tests ( χ2 ) or ANOVA, depending on the type of variable measure, always with 95% of Confidence, or P-Value ≤ 0,05. In the characterization of the Groups, the tests were undertaken with the values identified at the beginning of the treatment. Thus, the efficiency of the initiatives undertaken could be perceived. The objective was to identify the significant statistical differences, between the initial and final results of the tests.

The 10 CBT sessions were based on the previous study (King et al, 2007a), with some modifications and adaptations appropriate to the characteristics of the sample of the patients under study. The content of the sessions were distributed in the following way: PD education (including the educational concepts of anxiety, agoraphobia, panic, hyperventilation, respiratory re-education exercises (RR exercises), progressive muscular relaxation exercises (PMR exercises), preparation of a scale of "patient fears" from the smallest to greatest to cause anxiety, identification of cognitive distortions, cognitive restructuring (CR), symptom induction exercises (SIE), IE, IVE, reinforcement of conquests, observation of the difficulties in the procedures and maintenance of treatment gains.

The patients were encouraged to apply cognitive strategies at home, such as expose themselves to changes of temperature, physical exercise, amongst others, several times, with the purpose of inducing and tolerating the sensations with no therapeutic assistance.

The learning in the first phase of the treatment that BS related to panic are not really dangerous is essential to overcoming of agoraphobia and for the control of panic.

Standard model of the 10 CBT sessions:

1. st. Session: Education concerning the trajectory of PD and the preparation of a priority list of feared situations by the patient. Instructions to the patient of relaxation techniques, repeated whenever necessary. RR exercise: Placing ones hand above ones stomach, feeling the air passing through the diaphragm, perception of the abdominal movement at each respiration. Slow inspiration through the nose counting up to three, holding the respiration, counting up to three, and releasing the air slowly through the mouth counting up to six. Repetition of the exercise several times in a row. In continuity, Progressive Muscular Relaxation (PMR) (Jacobson, 1938) is undertaken with the individual, whereby the instructor seeks to exercise by tensioning four Groups of muscles for ten seconds and immediately after relaxing for another ten seconds. The latter are: 1st face; 2nd arms, shoulders, chest and neck; 3rd abdomen, spine, genital organs and 4th legs and feet.
2. nd. Session: explanation concerning the physiological mechanism of "fight and flight" (Barlow, 1988b), verification of the similarity between the sensation originating from this mechanism, compared with BS that emerge from panic. Undertake RR exercise, used constantly during the sessions. When one manages to alter the thoughts referring to the capacity to deal with feared situations, one is capable of controlling the physical symptoms.
3. rd. Session: model of hyperventilation that delineated by the rhythm and depth of the exaggerated respiration for the needs of the body at a specific given moment. The latter was undertaken with a patient sitting in a position of SIE hyperventilation: patient inspires and expires deeply for 90 seconds, observation of patient reactions and explanation of the reason for the emerging symptoms. Undertaking of RR exercise. The patient should understand that anticipated anxiety is characterized by anticipated thought processes, generally negative, of feared situations. Even in a secure situation if the mind interprets it as insecure, the body will react with a message of danger producing symptoms.
4. th. Session: SIE: -sitting, look fixedly at a light for a minute and afterwards standing up quickly and trying to read something. Analysis with the patient of the sensations present and the levels of negative, catastrophic and repetitive thoughts that have occurred. The patient begins to understand the origin of the symptoms and to perceive that they are inoffensive, learning to deal with them. In continuity, RR exercise is administered.
5. th. Session: explanation of the concepts of BS that can be accentuated due to a situation or to substances. Examples: exercising oneself or moving oneself quickly, brusque changes of temperature, bright light, use of caffeine, alcohol, medicines and irregular levels of respiration. Panic has it root in the fear of physical sensations (Rangé, 2001b).

   A patient was submitted to SIE: turning around in circles for a minute, afterwards stopping, understanding and giving a new positive significance to the reactions verified.

   Immediately after, RR exercise is administered.
6. th. Session: in PA some of the patient complaints were: ex: "I cannot breathe", or "I am going to suffocate". It was explained that it is natural to breathe excessively when one is anxious. The body seeks more energy in the form of oxygen to prepare itself to deal with danger. When the oxygen is not used in the same proportion in which it is consumed, the result is hyperventilation. The concepts of hyperventilation are remembered and SIE of the 4th session is repeated, followed by RR exercise.
7. th. Session: education concerning CR - The way events are interpreted is what determines the nature of the resulting emotional reactions (Rangé, 2001c). The patient should try to identify and give a new significance to the specific badly-adapted cognations. The concepts of Anticipated Anxiety (AA) and agoraphobic avoidance (PA-aa) (Beck, 1994) were clarified. Patients have the custom of myths in relation to PA: "I think I am going to lose control", "I think I am going to die", "I think I am going to have a heart attack", I think I am going mad", amongst others. The patient is instructed to question and contest his or her conjectures and beliefs concentrating on the realistic probabilities and gather evidence and forms to deal with the events.
8. th.Session: The IE refers to the fear learnt of internal state. Certain sensations of terror, similar to fear previously experienced, have the custom of indicating new possible PA (Muotri et al, 2007c). The automatic stimulus generated intensifies the feared sensations, creating a vicious circle. Undertake two SIE: Sitting down, place the patient's head between his or her legs for 30 seconds, afterwards sit up quickly and look to the ceiling. And other exercise: the patient holds his or her respiration until it can no longer be held while turning round in circles for 30 seconds. In continuity, analysis of the symptoms and trying to understand the originating causes. RR exercise is undertaken.
9. th. Session: Undertake three SIE: repeat the exercise of the 5th session and the two of the 8th session with subsequent administration of RR exercise. The purpose being for the individual to associate the symptom with the cause, explain that the symptoms emerge from physiological alterations triggered for some reason, differently from what one thought that BS emerged from nowhere, with no apparent reason. Previously, the patient would make a distorted association of the facts, interpreting tachycardia, perspiration, lack of breath, among others, as a sign of imminent death or loss of control and not as resulting from specific triggering factors.
10. th. Session: one SIE: the patient standing up turns his or her head from one side to the other for 30 seconds, stops and tries to fix his or her eyes on a spot on the wall. Repeat this exercise after SIE of the 3rd session, in continuity; recover the patient's physical balance and respiration with RR or PMR exercises. Evaluate the IVE concept regarding confronting the patient with agoraphobic situations or locations. Explain that agoraphobia is maintained by the fear of panicking or the experience of certain BS.

Real confrontation with the feared situation is repeated with each item of the priority list of the patient's fears, beginning with the least anxiety provocative, until reaching the most feared. Ask the patient to practise IVE whenever there is an opportunity.

Review the IVEs undertaken, encourage the practical repetitions, and discuss the difficulties in the procedures. The behaviour of exceeding oneself should be encouraged instead of unnecessary over precautions. Remind the patient that to run away from the IVE reinforces the maintenance of fear. The therapist stimulates thoughts concerning the avoided tasks and helps the patient with CR. The fact that the additional diagnostics have the tendency to decline after PD treatment should be commented. Ex: comorbidities such as depression, generalized anxiety and social phobia. Reaffirm that the fear response is inoffensive, passing and controllable, the BS appear and disappear, without the need of being avoided.

After the end of all the stages of the research, the two Groups were re-evaluated with same initial instruments. The Groups were compared, observing the changes that had occurred, the benefits, the losses and differences that had occurred because Group 1 had received accompaniment with CBT and medication, compared to Group 2 control that had only made use of medication with no CBT.

ELIGIBILITY:
Inclusion Criteria:

* The criteria for inclusion in the research was patients over 18 years old of both sexes with a diagnosis of PDA, with no serious comorbidities.

Exclusion Criteria:

* The patients that presented alcohol or drug dependency, mental retardation or serious mental disorders were excluded from the research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-05; Primary Completion 2006-08 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Number of panic attacks | 3 months

SECONDARY OUTCOMES:
Decrease agoraphobic symptoms | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio E Nardi, MD, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Institute of Psychiatry - UFRJ, Rio de Janeiro, Rio de Janeiro, Brazil